CLINICAL TRIAL: NCT05318911
Title: Antithrombotic Activities of a Novel Yogurt Drink: a Dietary Intervention Study
Brief Title: Antithrombotic Activities of a Novel Yogurt Drink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, Ioannis Zabetakis, Head of Department of Biological Sciences, University of Limerick
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2022_01_01_S&E
Record Dates: First submitted 2022-03-04; First posted 2022-04-08 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement Group (Active Comparator): 10 participants will provide baseline blood samples after overnight fasting, on day 0 of the study. Following this they will initially consume 200 mL of novel yogurt drink per day for a period of 28 days.
  Then, after a 2-week washout period in which the subjects do not take any yoghurt drink , Phase II of the clinical trial will commence. This is the crossover phase in which subjects who took YD will now be given a placebo drink, and vice versa, over 4 weeks. A total of 80 blood samples will be collected for analysis.
  Interventions: Dietary Supplement: Novel yogurt drink
- Placebo Group (Placebo Comparator): 10 participants will provide baseline blood samples after overnight fasting, on day 0 of the study. Following this they will initially consume 200 mL of placebo drink per day for a period of 28 days.
  Then, after a 2-week washout period in which the subjects do not take any placebo drink , Phase II of the clinical trial will commence. This is the crossover phase in which subjects who took YD will now be given a placebo drink, and vice versa, over 4 weeks. A total of 80 blood samples will be collected for analysis.
  Interventions: Other: Placebo Drink

INTERVENTIONS:
Dietary Supplement: Novel yogurt drink — Novel ovine yogurt drink containing polar lipids
  Arms: Supplement Group
Other: Placebo Drink — Placebo drink (skimmed milk)
  Arms: Placebo Group

SUMMARY:
This study aims to evaluate antithrombotic activities of novel yoghurt drink in healthy adult volunteers

DETAILED DESCRIPTION:
This randomized controlled, double-blinded crossover study aims to investigate the antithrombotic activities of a novel yoghurt drink in healthy adult volunteers. It is anticipated that the novel drink containing beneficial polar lipids will reduce platelet aggregation in participants and consequently decrease the onset of cardiovascular disease.

In Phase I, the subjects will provide blood samples after overnight fasting and then take either a yoghurt drink (YD) or placebo (that does not contain polar lipids) daily for 4 weeks. Following this period, they will again provide blood samples. Then, after a 2-week washout period in which the subjects do not take any yoghurt or placebo drink , Phase II of the clinical trial will commence. This is the crossover phase in which subjects who took YD will now be given a placebo drink, and vice versa, over 4 weeks. A total of 80 blood samples will be collected for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Volunteers need to be off medication and off any dietary supplements.
* Subjects must not have any blood clotting disorders or dyslipidaemia.
* Dairy intake needs to be within a normal range of 1-2 portions a week.
* Unwilling to follow the study requirements.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation of PRP samples in the presence of PAF | Participants' platelet activity will be assessed for up to roughly 6 months through study completion
  Platelet aggregation of participants' platelet-rich plasma samples (PRP) in the presence of the platelet agonist PAF will be assessed, using EC50 as a parameter.
Screening of plasma levels of cholesterol ( PL, LDL, HDL, VLDL). | The outcomes of this testing will be assessed for up to roughly 6 months through study completion.
  Platelet-rich plasma (PRP) levels of cholesterol ( PL, LDL, HDL, VLDL levels) will be assessed.
Screening plasma levels of inflammatory markers. | The outcomes of this testing will be assessed for up to roughly 6 months through study completion.
  Platelet-rich plasma levels of the inflammatory markers (IL-6, CRP. TNF-α, VEGF, VCAM-1 and PAFR) will all be screened.
Screening plasma levels of triglycerides. | The outcomes of this testing will be assessed for up to roughly 6 months through study completion.
  PRP levels of triglycerides will also be screened.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tsoupras A, Zabetakis I, Lordan R. Platelet aggregometry assay for evaluating the effects of platelet agonists and antiplatelet compounds on platelet function in vitro. MethodsX. 2018 Dec 26;6:63-70. doi: 10.1016/j.mex.2018.12.012. eCollection 2019. PMID 30619728